CLINICAL TRIAL: NCT01881009
Title: Nocturnal Closed-Loop Control Using An ePID (Enhanced Proportional Integral Derivative) Algorithm On An Android Platform With Remote Monitoring In A Closely Monitored Camp Setting: The OCL Camp Study
Brief Title: Medtronic Minimed Overnight Closed-Loop System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce A. Buckingham (Other)
Responsible Party: Sponsor-Investigator, Bruce A. Buckingham, MD, Professor, Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G130115 IRB 27462
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes Mellitus; Autoimmune Diabetes; Juvenile-Onset Diabetes; Diabetes, Mellitus, Type 1
Keywords: Diabetes; Insulin; Closed loop; Nocturnal glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient overnight (Experimental): Participants in this group will have an overnight evaluation to test safety of the closed-loop system therapy device.
  Interventions: Device: Hybrid Closed-loop System
- Summer Camp Session (Experimental): Participants in this group will receive either the sensor augmented pump or the close loop controller on the first night, then alternated treatment type each night for the duration of the study.
  Interventions: Device: Hybrid Closed-loop System; Device: Sensor-augmented pump

INTERVENTIONS:
Device: Hybrid Closed-loop System — Medtronic Revel insulin pump, Enlite 3 sensor, Minimed transmitter, PID-IFB (proportional-integral-derivative based with insulin feedback) algorithm on an Android platform with remote monitoring.
Device: Sensor-augmented pump — Medtronic Revel insulin pump, Enlite 3 sensor, Minimed transmitter.
  Arms: Summer Camp Session

SUMMARY:
To test the function and safety of the Medtronic Overnight Closed Loop (OCL) System in a closely monitored 12 hour overnight inpatient study. Once the safety of the device has been validated we will move the study to an outpatient diabetes camp setting. The camp setting will allow us to obtain pilot efficacy and safety data in a "real-life" environment.

We plan to compare the subject control nights to the subject nights on the OCL system to assess the percent of sensor glucose readings in the target range of 70-150 mg/dl. Based on previous research, we anticipate that the use of the OCL system will contribute to a greater percentage of sensor glucose readings in the target range.

DETAILED DESCRIPTION:
The steps are the same for the inpatient and camp studies, except that during the inpatient study subjects will have an IV inserted and blood samples will be obtained every 1/2 hour overnight. They will also have 20-30 minutes of activity in the afternoon and evening. After 16 subjects have entered the inpatient study, their data will be sent to the DSMB (Data Safety Monitoring Board) for review. If the studies show that these studies have met our predefined safety criteria, and the DSMB approves, we will then conduct our outpatient studies.

Step 1:

Subjects who are eligible for the study (camp or inpatient hospital) will be contacted by phone and email, the study will be explained to them, and after written consent is obtained, they will be enrolled in the study. They will be mailed a Bayer Next meter, control solutions, and glucose test strips.

Step 2: The will perform quality control test on the meter using the control solutions, and email these results to the study coordinator. For the week prior to the research center admission or camp they will be asked to use the Bayer meter to obtain two fasting glucose levels 20 minutes apart. They will be called by the study coordinator 3-5 days prior to admission to review these blood glucose testing requirements with the family. Subjects who have at least 3 days of data will be eligible for study participation.

Step 3: On arrival to the hospital, camp or bus stop subjects will bring an original informed consent signed by both parents and/or guardians if less than 18 years old. This generally occurs between 10 AM and noon at the camps, and we will have them arrive before lunch to the research center.

Step 4: The will have lunch, and within the first 3 hours after lunch (or within 3 hours of arrival to camp or the research center) they will have a history, limited physical exam and an A1c level and pregnancy test if female.

They will be assigned a unique 5 digit identifier: The first digit is for the camp session; the next two digits are for their cabin number; and the last two digits are for their subject ID (identification). Subject 30804 would be in camp session 3, assigned to cabin 8, and subject 4. All subjects enrolled will be assigned a subject ID which progressively increases across all camp sessions, i.e. during the summer there will be only one subject #4.

Step 5: Their Medtronic pump (from home) and Bayer meter will be uploaded. Two Enlite sensor will be used during the inpatient study. Only one Enlite sensor will be used during the camp phase of the study. All sensors will be inserted before 3pm and subjects will be given a study pump, and all their pump settings will be transferred to the study Revel 2.0 Medtronic Insulin Pump. They will receive training on the study pump and Enlite sensors. The CGM training will be done as a group session and will consist of the standard teaching which we developed for the JDRF (Juvenile Diabetes Research Foundation) randomized clinical trial. Insulin doses are only given by camp medical staff (including all correction doses), we will not use predictive alarms. Alarm thresholds will be set for 70 and 250 mg/dl during the day and on control nights. When the CLP is active at night, the local alarms on the Revel 2.0 pump will be turned off. There will be no rate of change alarms. There active insulin time will be set to 6 hours. This will probably be different from their usual setting, and this will be explained to that this setting is for safety purposes during this study. The bolus wizard feature of the pump will be turned on and used for all insulin doses. They may use the type of meal boluses they would routinely use for meals at home (standard and/or dual wave or square wave boluses).

Step 6: Data from their pump and meter download will be used to initialize the CLP. These initialization parameters will be entered into the Android phone assigned to them (which will remain with study staff). Their name will taped onto the phone, their study pump, home pump and meter using a labeler. The date and time will be entered into each device so they are all times are synchronized to the nearest minute.

Step 7: At camp they will be randomized by cabins, so that an equal number of campers will be assigned to have active closed-loop control on the first night or be in the control arm on the first night. Thereafter campers in each arm will alternate between receiving closed and open loop intervention nights.

Step 8: The Enlite sensor(s) will be calibrated 2 hours after insertion, before dinner and at 9 PM if there are no rate of change arrows at these times on the first day. Thereafter calibration values will be entered before meals and before the 9 PM snack if there are no rate of change arrows. These finger sticks are done under supervision of a counselor who makes sure that their hands are either washed or the finger is cleaned with alcohol and allowed to dry before the finger prick.

Step 9: At camp there will be evening activities after dinner, which can range from "capture-the-flag", scavenger hunts, dances, campfires, and other activities. During the inpatient hospital stay we will have some activity after dinner between 7-8 PM where subjects will wear a heart rate monitor with the goal of achieving an elevated heart rate which varies between 100 to 140 bpm for 20 - 30 minutes. This may be accomplished using an exercise treadmill or bicycle, or other aerobic activities (jumping jacks, stair climbing, brief sprints, etc.). The goal is to have some evening activities that mimic some of the variable activities that occur at camp, so that they are not sedentary after dinner.

Step 11: On arrival to their cabins after evening activities those assigned to closed-loop control will have their CLP systems activated. In the hospital this will begin at 9 PM.

1. The OCL system parameters on the Android controller are set to the values listed on the subject-specific OCL parameter document. These are verified by two study personnel cross-checking each other.
2. A fingerstick glucose will be obtained and entered into the CLP. The meter glucose must be between 70 to 350 mg/dl for the OCL to be activated. At the same time a serum ketone test will be obtained with a Precision Xtra meter or a NovaStat meter and the serum ketones must be ≤ 0.6 mmol/L to proceed with the study.
3. The Translator, Revel 2.0 Insulin Pump and MiniLink must be within 6 feet of each other. The OCL controller (on Android platform) will be in the subject/campers room/cabin but they will not have direct contact with the controller.
4. The OCL will be activated. The system may not activate if the sensor and meter glucose readings show a greater than 20% difference. In this case the threshold alarms on the pump will be activated at 70 and 250 mg/dl and the OCL will not be used.

Step 12: The CLP (Closed Loop Platform, Android phone) will establish communication with the intranet at camp and remote monitoring will be confirmed by viewing data on a iPAD connected to the camp intranet. In the hospital CLP will establish communication with the hospital intranet service, and remote monitoring will be confirmed on a computer outside the patients room and on an iPAD.

Step 14: Patient management decisions based on meter glucose readings (and possible ketone readings during the study).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a subject must meet the following criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and a Medtronic insulin infusion pump for at least 3 months The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
* Age 10.0 - 35 years

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

* Diabetic ketoacidosis in the past month
* Hypoglycemic seizure or loss of consciousness in the past 3 months
* History of seizure disorder (except for hypoglycemic seizure)
* History of any heart disease including coronary artery disease, heart failure, or arrhythmias
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria).
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal disorder
  * Abuse of alcohol
* Pregnancy

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08-03 (Actual); Study Completion 2013-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ly TT, Keenan DB, Roy A, Han J, Grosman B, Cantwell M, Kurtz N, von Eyben R, Clinton P, Wilson DM, Buckingham BA. Automated Overnight Closed-Loop Control Using a Proportional-Integral-Derivative Algorithm with Insulin Feedback in Children and Adolescents with Type 1 Diabetes at Diabetes Camp. Diabetes Technol Ther. 2016 Jun;18(6):377-84. doi: 10.1089/dia.2015.0431. Epub 2016 May 16. PMID 27183197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment included mailing/emailing/calling to the families who registered the camp sessions when this study was conducted. Other sources of recruitment included chart review, Stanford Peds Endo Facebook page, Stanford Peds Endo website, support groups, department newsletter, clinic visits, and group visits.
Groups:
- Inpatient Overnight: Overnight evaluation to test safety of the closed-loop system therapy device.
- Summer Camp Session: Participants were considered to be a single group, receiving the same interventions, either the sensor augmented pump or the close loop controller on the first night, then alternated treatment type each night for the duration of the study. The sensor augmented pump was considered to be the control.
Period: Inpatient Safety Testing (22 Hours)
Arm/Group | Inpatient Overnight | Summer Camp Session
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Summer Camp Session (6 Days)
Arm/Group | Inpatient Overnight | Summer Camp Session
Started | 0 | 22
Completed | 0 | 21
Not Completed | 0 | 1
Not completed — Unable to wear device | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant who withdrew from the summer camp session was excluded from the analysis.
Groups:
- Summer Camp Session: Participants were considered to be a single group, receiving the same interventions, either the sensor augmented pump or the close loop controller on the first night, then alternated treatment type each night for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Inpatient Overnight | Summer Camp Session | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 19 | 33
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (2.5) | 14.7 (3.9) | 14.95 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 20 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Target Sensor Glucose 70-150 mg/dl
Description: Compared to control nights, the percent of time in the target range of 70-150 mg/dl according to sensor glucose readings.
Time Frame: Approximately 12 hours
Population: Intention to treat analysis of the summer camp session. 1 participant who withdrew from the summer camp session was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage of time
Units Other Than Participants: Nights analyzed (all participants)
Groups:
- Closed Loop Nights: Data for nights that participants received closed loop controller treatment.
- Control Nights: Data for nights that participants received sensor augmented pump treatment.
Arm/Group | Closed Loop Nights | Control Nights
Number analyzed (Participants) | 21 | 21
Number analyzed (Nights analyzed (all participants)) | 55 | 52
percentage of time | 66.4 (4.2) | 50.6 (4.3)
Statistical Analysis 1: Comparison: Closed Loop Nights vs Control Nights; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Target Sensor Glucose 70-180 mg/dl
Description: Compared to control nights, the percent of time in the target range of 70-180 mg/dl according to sensor glucose readings.
Time Frame: Approximately 12 hours
Population: Target sensor glucose 70-180 mb/dl was a secondary outcome for the summer camp group only. 1 participant who withdrew from the summer camp session was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage of time
Units Other Than Participants: Nights analyzed (all participants)
Arm/Group | Closed Loop Nights | Control Nights
Number analyzed (Participants) | 21 | 21
Number analyzed (Nights analyzed (all participants)) | 55 | 52
percentage of time | 79.9 (3.8) | 60.0 (4.0)
Statistical Analysis 1: Comparison: Closed Loop Nights vs Control Nights; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Target Sensor Glucose 70-150 mg/dl
Description: Percent of time in the target range of 70-150 mg/dl according to sensor glucose readings.
Time Frame: Approximately 12 hours
Population: Intention to treat analysis of the inpatient overnight group. 3 participants that did not complete the inpatient overnight are excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Nights analyzed (all participants)
Arm/Group | Inpatient Overnight
Number analyzed (Participants) | 13
Number analyzed (Nights analyzed (all participants)) | 13
percentage of time | 63 [41 to 89]

ADVERSE EVENTS:
Time Frame: On-study adverse events were collected for 22 hours in the Inpatient Overnight group, and for 6 days in the Summer Camp Session group.
Arm/Group | Inpatient Overnight | Summer Camp Session
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/22
Other Adverse Events (participants affected / at risk) | 0/16 | 21/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Overnight (N=16) | Summer Camp Session (N=22)
Hypoglycemia and hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No